CLINICAL TRIAL: NCT00965302
Title: Sleeve Gastrectomy vs Medical Management for Remission of Diabetes in Mild to Moderately Obese Patients
Brief Title: Sleeve Gastrectomy Versus Medical Management for Remission of Diabetes in Mild to Moderately Obese Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator did not submit an annual continuation report with the Institutional Review Board and the study was officially removed from IRB regulatory oversight on Sep 2014, based on 32 CFR 219.109e. The study officially expired/terminated.
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Responsible Party: Jason M. Pfluke, MD MAJ USAF MC, Wilford Hall Medical Center, United States Air Force
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWH20090068H
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: Obesity; Diabetes mellitus, Type 2; Sleeve gastrectomy; Metabolic surgery
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive medical management of Type 2 DM (Active Comparator): Intensive medical management of Type II diabetes will include visits every three months for a year with an endocrinologist, with lifestyle counseling, weight management, regular exercise, and glucose control forming the core of the medical therapy.
  Interventions: Behavioral: Intensive medical management
- Laparoscopic sleeve gastrectomy (Experimental): Laparoscopic sleeve gastrectomy is performed as part of a bariatric surgical program emphasizing healthy dietary choices, regular exercise, and glucose control.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Laparoscopic sleeve gastrectomy, also known as vertical sleeve gastrectomy, sleeve gastroplasty, or sleeve gastrectomy, will be performed over a 32 to 40 French sizing bougie.
  Arms: Laparoscopic sleeve gastrectomy
Behavioral: Intensive medical management — Intensive medical therapy for Diabetes mellitus, Type 2, will include weight management counseling, exercise, glucose control, and healthy dietary choices.
  Arms: Intensive medical management of Type 2 DM

SUMMARY:
The investigators plan to randomize mild to moderately obese (BMI 30-34.9) subjects to medical management (diet, exercise, and best medical therapy) versus sleeve gastrectomy with medical management, with a primary endpoint of diabetes remission (normal fasting glucose, off medications and insulin) at one year. Sleeve gastrectomy (also called greater curvature gastrectomy, vertical sleeve gastrectomy, and sleeve gastroplasty) involves stapled resection of the gastric fundus. Secondary endpoints include weight loss, improvement in hypertension, sleep apnea, c-reactive protein, and fasting lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus, Type 2
* Body Mass Index (BMI) 30-34.9
* Able to understand and comply with study process

Exclusion Criteria:

* Pregnancy
* Prior bariatric surgery
* Diabetes mellitus, Type 1
* Renal impairment
* Cirrhosis or portal hypertension
* Diabetes secondary to a specific condition
* Recent internal malignancy (<5 years)
* Recent major vascular event
* Drug or alcohol dependence
* Uncontrolled psychiatric disease
* Crippling cardiopulmonary disease
* Prohibitive anatomic features (extensive prior surgery, giant paraesophageal hernia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-08; Primary Completion 2012-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Diabetes remission | 1 year

SECONDARY OUTCOMES:
Weight loss | 1 year
Obstructive sleep apnea remission | 1 year
Fasting lipid profile | 1 year
c-reactive protein | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Pfluke, MD, Principal Investigator — Wilford Hall Medical Center, United States Air Force
Locations (1):
- Wilford Hall Medical Center, San Antonio, Texas, United States

REFERENCES:
- [Background] O'Brien PE, Dixon JB, Laurie C, Skinner S, Proietto J, McNeil J, Strauss B, Marks S, Schachter L, Chapman L, Anderson M. Treatment of mild to moderate obesity with laparoscopic adjustable gastric banding or an intensive medical program: a randomized trial. Ann Intern Med. 2006 May 2;144(9):625-33. doi: 10.7326/0003-4819-144-9-200605020-00005. PMID 16670131
- [Background] Kakoulidis TP, Karringer A, Gloaguen T, Arvidsson D. Initial results with sleeve gastrectomy for patients with class I obesity (BMI 30-35 kg/m2). Surg Obes Relat Dis. 2009 Jul-Aug;5(4):425-8. doi: 10.1016/j.soard.2008.09.009. Epub 2008 Sep 26. PMID 18996758
- [Background] Lee CM, Cirangle PT, Jossart GH. Vertical gastrectomy for morbid obesity in 216 patients: report of two-year results. Surg Endosc. 2007 Oct;21(10):1810-6. doi: 10.1007/s00464-007-9276-y. Epub 2007 Mar 14. PMID 17356932
- [Background] Dixon JB, O'Brien PE, Playfair J, Chapman L, Schachter LM, Skinner S, Proietto J, Bailey M, Anderson M. Adjustable gastric banding and conventional therapy for type 2 diabetes: a randomized controlled trial. JAMA. 2008 Jan 23;299(3):316-23. doi: 10.1001/jama.299.3.316. PMID 18212316
- [Background] Cohen R, Pinheiro JS, Correa JL, Schiavon CA. Laparoscopic Roux-en-Y gastric bypass for BMI < 35 kg/m(2): a tailored approach. Surg Obes Relat Dis. 2006 May-Jun;2(3):401-4, discussion 404. doi: 10.1016/j.soard.2006.02.011. PMID 16925363